CLINICAL TRIAL: NCT06664853
Title: An Open-Label Extension Study of EryDex in Patients With Ataxia Telangiectasia Following Participation in Study IEDAT-04-2022 (NEAT)
Brief Title: Open-Label Extension of EryDex Study IEDAT-04-2022
Acronym: OLE_NEAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEDAT-05-2024
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ataxia Telangiectasia
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexamethasone sodium phosphate (Experimental): intravenous (IV) infusion of dexamethasone sodium phosphate (DSP) encapsulated in autologous erythrocytes using the EryDex System (EDS)
  Interventions: Drug: Dexamethasone sodium phosphate

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate — Dexamethasone Sodium Phosphate encapsulated in autologous erythrocytes and administered via intravenous (IV) infusion

SUMMARY:
This is an international, multi-center, prospective, open-label, non-comparative study to provide EryDex treatment to ataxia telangiectasia (A-T) patients who complete the IEDAT-04-2022 trial on the neurological effects of EryDex on subjects with ataxia telangiectasia (NEAT trial).

DETAILED DESCRIPTION:
The IEDAT-05-2024 study aims to provide EryDex (dexamethasone sodium phosphate encapsulated into autologous erythrocytes) treatment to patients who complete the full study treatment period (including those receiving placebo) in the IEDAT-04-2022 (NEAT) study, who complete the study assessments, do not present safety contraindications to continuation of treatment, and provide informed consent. The open-label extension (OLE) treatment period will be 12 months. Participants will be considered to have completed the study when Visit 14 (Safety Follow-up) has been performed.

ELIGIBILITY:
Inclusion Criteria:

* body weight ≥15 kg
* participation in IEDAT-04-2022 study and its completion, including final efficacy and safety assessments

Exclusion Criteria:

* safety contraindications for continuation of treatment, as determined by the investigator
* clinically significant immune impairment that, in the opinion of the Investigator, precludes further treatment with corticosteroids
* Current neoplastic disease or previous neoplastic disease not in remission for at least 2 years.
* requiring treatment with a systemic corticosteroid

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | through study completion, up to 14 months
  Number of patients presenting at least one treatment emergent adverse event (TEAE)
Incidence of treatment emergent adverse events leading to intervention discontinuation | through study completion, up to 14 months
  Number of patients presenting at least one treatment emergent adverse event (TEAE) leading to intervention discontinuation
Incidence of serious adverse events | through study completion, up to 14 months
  Number of patients presenting at least one serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Thye, MD, Study Director — Quince Therapeutics S.p.A.
Locations (22):
- United States (6):
  - University of California Los Angeles (UCLA), Ataxia Center and HD Center of excellence, Los Angeles, California
  - The Johns Hopkins Hospital, Division of pediatric allergy and immunology, Baltimore, Maryland
  - Saint Peter's University Hospital, Inc., New Brunswick, New Jersey
  - Biotrial Inc., Newark, New Jersey
  - Cincinnati Children's Hospital, Division of neurology, Cincinnati, Ohio
  - UT Health Houston, Department of pediatrics, division of child & adolescent neurology, Houston, Texas
- Copenhagen University Hospital, Rigshospitalet, Department of Pediatric Neurology, Copenhagen, Denmark
- Germany (2):
  - IKF Pneumologie GmbH & Co. KG; Institut für klinische Forschung Pneumologie Clinical Research Center Respiratory Diseases, Frankfurt am Main, Hesse
  - University Hospital Frankfurt, Pediatric and Adolescent Clinic, Frankfurt
- Italy (2):
  - Spedali Civili di Brescia, Pediatric immunology department, Brescia
  - Policlinico Umberto I, La sapienza University, Department of neurosciences and menthal health, Roma
- Oslo University Hospital, Rikshospitalet, Division of Pediatric and Adolescent Medicine, Norwegian National Unit for Newborn Screening, Oslo, Norway
- Poland (2):
  - MedPolonia sp zoo, Poznan
  - Instytut "Pomnik-Centrum Zdrowia Dziecka", Immunology clinic, Warsaw
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Department of pediatric neurology, Barcelona
  - Hospital Universitario La Paz, Department of pediatric neurology, Madrid
  - Universitary Hospital Virgen del Rocío, Seville
- University Children's Hospital Zürich - Eleonore Foundation, Zurich, Switzerland
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - St George's University Hospitals NHS Foundation Trust, Centre for Neonatal and Paediatric Infection, London
  - Great Ormond Street Hospital for Children, Zayed Centre for Research, London
  - Nottingham Children's Hospital, Queen's Medical Center, Children's neurology, Nottingham

IPD SHARING:
Plan to Share IPD: No